CLINICAL TRIAL: NCT03752112
Title: Trial Evaluating the Clinical Efficacy of Cefixime for Treatment of Early Syphilis in Non-pregnant Women
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: World Health Organization (Other)
Responsible Party: Principal Investigator, Melanie Taylor, Medical Offier, World Health Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC0003096
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Syphilis Female
Keywords: Syphilis; Women; Cefixime; Brazil; Sexually Transmitted Infection; STI
MeSH Terms: conditions — Syphilis; Sexually Transmitted Diseases | interventions — Cefixime; Methods

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2 trial to evaluate the efficacy and safety of cefixime for use in treating women with acute syphilis.
  This is a randomized, non-comparative, open label study assessing the efficacy and safety of cefixime 400mg taken orally two times a day for 10 consecutive days in non-pregnant women with early syphilis infection.To benchmark the performance of benzathine penicillin in the study population being used for cefixime, The investigators will include a contemporary arm of participants that will receive standard of care treatment with benzathine penicillin according to the Brazil national STI treatment guidelines. The investigators will use a ratio of 2 patients receiving cefixime to 1 patient receiving benzathine penicillin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cefixime (Experimental): cefixime 400mg taken orally two times a day for 10 consecutive days in non-pregnant women with early syphilis infection.
  Interventions: Drug: Cefixime
- Benzathine penicillin (Other): To benchmark the performance of benzathine penicillin in the study population being used for cefixime, the investigators will include a contemporary arm of participants that will receive standard of care treatment with benzathine penicillin according to the Brazil national STI treatment guidelines. The investigators will use a ratio of 2 patients receiving cefixime to 1 patient receiving benzathine penicillin.
  Interventions: Drug: Benzathine penicillin 2.4 million units

INTERVENTIONS:
Drug: Cefixime — Cefixime 400mg taken orally two times a day for 10 consecutive days in non-pregnant women with early syphilis infection
  Other Names: Intervention
  Arms: Cefixime
Drug: Benzathine penicillin 2.4 million units — Benzathine penicillin 2.4 million units: The investigators will include a contemporary arm of participants that will receive standard of care treatment with Benzathine penicillin 2.4 million units according to the Brazil national STI treatment guidelines. The investigators will use a ratio of 2 patients receiving cefixime to 1 patient receiving benzathine penicillin.This non-comparator arm of benzathine penicillin will be included to account for study population differences in terms of stage of disease, history of prior infection, experience of re-infection, experience of serofast state, or other co-factors that could impact serological response
  Other Names: Standard treatment
  Arms: Benzathine penicillin

SUMMARY:
Hypotheses The antibiotic, Cefixime, for use in non-pregnant women with early syphilis will be efficacious and safe.

Primary Objective The primary objective of the study is to demonstrate the efficacy, as measured by a 4 fold decrease in Rapid Plasma Reagin (RPR) titer from baseline to 6 months after treatment, with Cefixime 400mg taken orally two times a day for 10 consecutive days.

Secondary Objective The secondary objective of the study is to determine the safety, as measured by the number of grade 3 or greater toxicities experienced, using the NIH/NCI toxicity score, during or after treatment with Cefixime 400mg taken orally two times a day for 10 consecutive days.

DETAILED DESCRIPTION:
Hypotheses The antibiotic, Cefixime, for use in non-pregnant women with early syphilis will be efficacious and safe.

Primary Objective The primary objective of the study is to demonstrate the efficacy, as measured by a 4 fold decrease in Rapid Plasma Reagin (RPR) titer from baseline to 6 months after treatment, with Cefixime 400mg taken orally two times a day for 10 consecutive days.

Secondary Objective The secondary objective of the study is to determine the safety, as measured by the number of grade 3 or greater toxicities experienced, using the NIH/NCI toxicity score (10), during or after treatment with Cefixime 400mg taken orally two times a day for 10 consecutive days.

Methods Study design This is a randomized, non-comparative, open-label study assessing the efficacy and safety of cefixime 400mg taken orally two times a day for 10 consecutive days in non-pregnant women with early syphilis infection.

Study population and enrolment sites Numerous regions of Brazil have experienced increases in syphilis diagnoses during the previous 5 years The study sites were chosen from three cities in three separate regions (states) of Brazil based on: (1) increases in syphilis case reports, (2) access to clinics where patients are screened and treated for syphilis; (3) willingness of clinic sites and staff to participate in this research, and (4) the availability of experienced researchers with experience in studying syphilis to serve as co-investigators.

The study population will include non-pregnant women (ages 18 and over) diagnosed with early syphilis (RPR titers >1:8) recruited from 7 clinics in three cities from three states in Brazil. These include: (1) Three clinics in the city of Fortaleza (Ceara State), coordinated by the University of Fortaleza (UNIFOR): (a) Carlos Ribeiro, (a) Meireles, and (c) Federal University. Syphilis epidemiology for each site in Annex 1. (2) Two University ObGyn Clinics in the city of Pelotas (state of Rio Grande do Sul) (5-6 cases of syphilis/week) a) Ambulatorio de Ginecologia e Obstetrícia - Faculdade de Medicina - Universidade Federal de Pelotas and b) Ambulatorio de Ginecologia e Obstetrícia - Campus da Saúde - Universidade Católica de Pelotas; and (3) Two clinics in Vitoria (State of Espirito Santo): (1) Reference Center for Sexually Transmitted Diseases (http://www.vitoria.es.gov.br/cidadao/centro-de-referencia-em-infeccoes-sexualmente-transmissiveis). (2) Hospital Universitário Cassiano Antonio Moraes - UFES.

Patients identified during standard of care testing with a positive rapid syphilis test and an RPR titer of greater than or equal to 1:8 will be referred to the study and offered enrollment according to the following description.

Non-study clinic-site staff will perform the first screening rapid finger-stick test for syphilis. The rapid syphilis test currently used in these clinics detects both new (acute) infection and old treated infection but does not distinguish between the two. Patients that are positive for the syphilis rapid finger-stick test will be notified by non-study staff of this result and the need for additional testing using the RPR test according to standard of care. Blood will be collected for the confirmatory RPR test by non-study staff. These patients will be notified of RPR results in approximately 3 days to 1 week. The results a confirmed syphilis diagnosis and of the RPR test results for those patients that are eligible for enrolment in the study (RPR >1:8) will be provided by a study nurse. The study will be explained to eligible participants (RPR titer of >1:8) by this study nurse, and if women express interest in participating, informed consent will be obtained. It is expected that an enrolment visit could last approximately 1.5 hours.

Patients that are not eligible for the study (negative RPR or RPR with titer <1:8) will receive syphilis RPR results from non-study staff.

Pregnancy tests will be completed on all potential participants and those that test positive will not be enrolled in the study.

The timing of the recruitment process will depend on the number of women diagnosed with syphilis and who have an RPR titer >1:8 and who consent to participate in the study. It is anticipated that enrollment will take approximately 1 year to complete.

To benchmark the performance of benzathine penicillin in the study population being used for cefixime, The investigators will include a contemporary arm of participants that will receive standard of care treatment with benzathine penicillin according to the Brazil national sexually transmitted infection (STI) treatment guidelines. The investigators will use a ratio of 2 patients receiving cefixime to 1 patient receiving benzathine penicillin.

This non-comparator arm of benzathine penicillin will be included to account for study population differences in terms of stage of disease, history of prior infection, experience of re-infection, experience of serofast state, or other co-factors that could impact serological response. An estimate of performance of this standard of care will be calculated, but this will not be compared directly to the study intervention.

The investigators will enrol 180 eligible women into the study: 120 for the cefixime arm and 60 for the benzathine penicillin arm. It is anticipated that enrollment will take approximately 1 year to complete. Patients will be participating in the study for approximately 9 months. The study is expected to last for approximately two years. Women that are referred to the study but decline enrolment will be treated at the clinic following national STI treatment guidelines for syphilis.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 18 years of age or older
2. Non-pregnant
3. Able to provide informed consent
4. Test positive for syphilis with a positive TPPA AND an RPR titer equal to or greater than 1:8
5. Non-cephalosporin allergic
6. Non-penicillin allergic
7. Agree to be called once a day by study staff to be reminded to take study drug
8. Able to swallow pills
9. Willing to attend follow-up visits at 3, 6, and 9 months after completion of the study treatment
10. Willing to take oral contraceptive or use condom to prevent pregnancy during the study period
11. HIV negative

Exclusion Criteria:

1) Female under 18 years of age 2) HIV positive 3) Pregnancy test positive or clinical pregnancy 4) Prior history of syphilis or syphilis treatment within 6 months of study screening 5) Allergy to penicillin or cephalosporins (including allergy to cefixime) 6) In the judgment of the interviewer, has a medical condition or other factor that might affect their ability to follow the protocol 7) Previous enrollment in the study 8) Presenting a condition that would not allow reliable informed consent (alcohol abuse or substance misuse) 9) Lacking mental capacity to give informed consent to participation

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on biologic gender
Enrollment: 180 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative RPR titer change | 6 months following last dose of Cefixime 400 mg
  RPR titer response at 6 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE with cefixime | Daily after the first dose of cefixime 400mg orally through 10 days after the first dose
  Number of participants with treatment-related adverse events as assessed by CTCAE. Information on side effects will be collected daily for 10 days of administration of cefixime using a pre-established list of most commonly reported side effects and a grade scale will be applied using the Common Terminology Criteria for Adverse Events.
The number of participants reporting tolerability of cefixime | Daily after the first dose of cefixime 400mg orally through 10 days after the first dose and qualitative overall assessment of tolerability measured via questionnaire 14 days after the first dose of cefixime
  Tolerability: The number of participants reporting tolerability of cefixime as measured by quantitative reported experience of common side effects and qualitative experience of tolerance of the regimen as collected through daily questionnaires and an end treatment questionnaire at 14 days after the first dose of cefixime.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie M Taylor, MD, Principal Investigator — World Health Organization; Nathalie JN Broutet, MD, Study Director — World Health Organization; Edna O Kara, MD, Study Chair — World Health Organization
Locations (1):
- Fortaleza University, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Beginning 9 months and ending 24 months following article publication, the supporting information that will be shared for IPD are all data that underlie the results in the publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 24 months following article publication,
Access Criteria: * Access will be provided to investigators whose proposed use of data has been approved by an independent review committee identified for this purpose
  * Data whose goal is to achieve aims in the approved proposal
  * The way proposals should be submitted will be decided and informed after WHO standard operating procedure (in development) for this purpose is complete.

REFERENCES:
- [Background] Workowski KA, Bolan GA; Centers for Disease Control and Prevention. Sexually transmitted diseases treatment guidelines, 2015. MMWR Recomm Rep. 2015 Jun 5;64(RR-03):1-137. PMID 26042815
- [Background] WHO Guidelines for the Treatment of Treponema pallidum (Syphilis). Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK384904/ PMID 27631046
- [Background] Liang Z, Chen YP, Yang CS, Guo W, Jiang XX, Xu XF, Feng SX, Liu YQ, Jiang G. Meta-analysis of ceftriaxone compared with penicillin for the treatment of syphilis. Int J Antimicrob Agents. 2016 Jan;47(1):6-11. doi: 10.1016/j.ijantimicag.2015.10.020. Epub 2015 Nov 23. PMID 26724187
- [Background] Norris SJ, Cox DL, Weinstock GM. Biology of Treponema pallidum: correlation of functional activities with genome sequence data. J Mol Microbiol Biotechnol. 2001 Jan;3(1):37-62. PMID 11200228
- [Background] Faulkner RD, Fernandez P, Lawrence G, Sia LL, Falkowski AJ, Weiss AI, Yacobi A, Silber BM. Absolute bioavailability of cefixime in man. J Clin Pharmacol. 1988 Aug;28(8):700-6. doi: 10.1002/j.1552-4604.1988.tb03203.x. PMID 3216036
- [Background] Faulkner RD, Bohaychuk W, Haynes JD, Desjardins RE, Yacobi A, Silber BM. The pharmacokinetics of cefixime in the fasted and fed state. Eur J Clin Pharmacol. 1988;34(5):525-8. doi: 10.1007/BF01046715. PMID 3203716
- [Background] Barbee LA, Nayak SU, Blumer JL, O'Riordan MA, Gray W, Zenilman JM, Golden MR, Griffiss JM. A Phase 1 Pharmacokinetic and Safety Study of Extended-Duration, High-dose Cefixime for Cephalosporin-resistant Neisseria gonorrhoeae in the Pharynx. Sex Transm Dis. 2018 Oct;45(10):677-683. doi: 10.1097/OLQ.0000000000000844. PMID 29624558
- [Background] Rafal'skii VV, Dovgan' EV, Kozyrev IuV, Gustovarova TA, Khlybova SV, Novoselova AV, Filippenko NG, Likhikh DG. [The efficacy and safety of cefixime and amoxicillin/clavulanate in the treatment of asymptomatic bacteriuria in pregnant women: a randomized, prospective, multicenter study]. Urologiia. 2013 Sep-Oct;(5):24, 26-8. Russian. PMID 24437236
- [Background] Nurse-Findlay S, Taylor MM, Savage M, Mello MB, Saliyou S, Lavayen M, Seghers F, Campbell ML, Birgirimana F, Ouedraogo L, Newman Owiredu M, Kidula N, Pyne-Mercier L. Shortages of benzathine penicillin for prevention of mother-to-child transmission of syphilis: An evaluation from multi-country surveys and stakeholder interviews. PLoS Med. 2017 Dec 27;14(12):e1002473. doi: 10.1371/journal.pmed.1002473. eCollection 2017 Dec. PMID 29281619
- [Background] U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES. National Institutes of Health National Cancer Institute. Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 . https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03/Archive/CTCAE_4.0_2009-05-29_QuickReference_8.5x11.pdf
- [Background] Hook EW 3rd, Behets F, Van Damme K, Ravelomanana N, Leone P, Sena AC, Martin D, Langley C, McNeil L, Wolff M. A phase III equivalence trial of azithromycin versus benzathine penicillin for treatment of early syphilis. J Infect Dis. 2010 Jun 1;201(11):1729-35. doi: 10.1086/652239. PMID 20402591
- [Background] Cao Y, Su X, Wang Q, Xue H, Zhu X, Zhang C, Jiang J, Qi S, Gong X, Zhu X, Pan M, Ren H, Hu W, Wei Z, Tian M, Liu W. A Multicenter Study Evaluating Ceftriaxone and Benzathine Penicillin G as Treatment Agents for Early Syphilis in Jiangsu, China. Clin Infect Dis. 2017 Oct 30;65(10):1683-1688. doi: 10.1093/cid/cix611. PMID 29020150
- [Derived] Stafylis C, Keith K, Mehta S, Tellalian D, Burian P, Millner C, Klausner JD. Clinical Efficacy of Cefixime for the Treatment of Early Syphilis. Clin Infect Dis. 2021 Sep 7;73(5):907-910. doi: 10.1093/cid/ciab187. PMID 33640982
- [Derived] Taylor MM, Kara EO, Araujo MAL, Silveira MF, Miranda AE, Branco Coelho IC, Bazzo ML, Mendes Pereira GF, Pereira Giozza S, Bermudez XPD, Mello MB, Habib N, Nguyen MH, Thwin SS, Broutet N. Phase II trial evaluating the clinical efficacy of cefixime for treatment of active syphilis in non-pregnant women in Brazil (CeBra). BMC Infect Dis. 2020 Jun 10;20(1):405. doi: 10.1186/s12879-020-04980-1. PMID 32522244